CLINICAL TRIAL: NCT00183768
Title: Antidepressant Treatment to Reduce HIV Risk Among IDUs
Brief Title: Cognitive Behavioral Therapy Combined With Antidepressants to Reduce HIV Risk and Drug Relapse Among Depressed Intravenous Drug Users
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Michael Stein, M.D./Principal Investigator, RI Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH061141 (NIH); R01MH061141 (NIH); DAHBR AZ-M
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections; Depression; Substance-Related Disorders
Keywords: Cognitive Behavioral Treatment For Depression; Antidepressant Psychopharmacology; HIV Risk Behavior; Injection Drug Use
MeSH Terms: conditions — HIV Infections; Depression; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy; Psychopharmacology

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy
Behavioral: Psychopharmacology

SUMMARY:
This study will evaluate the effectiveness of combining cognitive behavioral therapy (CBT) and antidepressants in reducing HIV risk behavior and drug relapse rates in depressed intravenous drug users.

DETAILED DESCRIPTION:
Depression is common among injection drug users (IDUs); it is estimated that up to 50% of IDUs meet the diagnostic criteria for major depressive disorder, a severe form of depression. The combination of drug abuse and depression increases the likelihood of engaging in HIV high-risk behaviors such as unprotected sex and the use of unhygienic needles to inject drugs. Research has shown that IDUs who receive treatment for depression have lower rates of drug relapse and are less likely to engage in high-risk sexual behavior compared to IDUs who have not received treatment for depression. Combination treatment, which includes cognitive behavioral therapy (CBT) and antidepressant medication, has been shown to be the most effective treatment for depression. This study will evaluate the effectiveness of combination treatment in reducing HIV risk behaviors and drug relapse rates in cocaine or opiate addicted IDUs with a diagnosis of depression.

In this 9-month study, participants will be randomly assigned to either a combination treatment group or an assessment only group that will receive no treatment. Participants assigned to combination treatment will receive the antidepressant Celexa, and will attend 8 CBT sessions and 7 psychopharmacology sessions. Each CBT session will last about 60 minutes and each psychopharmacology session will last about 15 minutes. If a participant does not respond well to Celexa, Wellbutrin or Effexor may be taken instead. Participants in both groups will attend 4 study visits during which they will complete standardized psychological questionnaires and interviews to assess depression levels, drug use, and high-risk sexual behaviors. Blood will be drawn at baseline and Month 9 for HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for major depression, dysthymia, substance-induced major depression, or major depression plus dysthymia
* Score of greater than 14 on the Hamilton Depression Rating Scale
* Involved in HIV risk behaviors
* Current opiate or cocaine use
* Basic proficiency in English

Exclusion Criteria:

* Current suicidal risk or ideation
* Current psychotic symptoms
* Simultaneous medical disorder that might make psychopharmacological treatment medically inadvisable
* History of bipolar disorder, schizophrenia, schizo-affective disorder, schizophreniform disorder, or paranoid disorder
* Currently taking other medications for depression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 1999-09; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
HIV risk behavior; measured at Month 9

SECONDARY OUTCOMES:
Depression severity; measured at Month 9

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Rhode Island Hospital; Penelope Dennehy, MD, Study Director — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Stein MD, Herman DS, Solomon DA, Anthony JL, Anderson BJ, Ramsey SE, Miller IW. Adherence to treatment of depression in active injection drug users: the minerva study. J Subst Abuse Treat. 2004 Mar;26(2):87-93. doi: 10.1016/S0740-5472(03)00160-0. PMID 15050085
- [Result] Stein MD, Solomon DA, Herman DS, Anthony JL, Ramsey SE, Anderson BJ, Miller IW. Pharmacotherapy plus psychotherapy for treatment of depression in active injection drug users. Arch Gen Psychiatry. 2004 Feb;61(2):152-9. doi: 10.1001/archpsyc.61.2.152. PMID 14757591
- [Result] Stein MD, Solomon DA, Herman DS, Anderson BJ, Miller I. Depression severity and drug injection HIV risk behaviors. Am J Psychiatry. 2003 Sep;160(9):1659-62. doi: 10.1176/appi.ajp.160.9.1659. PMID 12944342